CLINICAL TRIAL: NCT00033540
Title: A Phase II Trial of Gemcitabine (NSC-613327) and Capecitabine (NSC-712807) in Patients With Unresectable or Metastatic Gallbladder or Cholangiocarcinoma
Brief Title: S0202 Gemcitabine and Capecitabine for Unresectable Locally Advanced Metastatic Gallbladder Cancer or Cholangiocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069299; S0202 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Results first posted 2012-08-28 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-08

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer
Keywords: unresectable gallbladder cancer; recurrent gallbladder cancer; unresectable extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; adenocarcinoma of the gallbladder; adenocarcinoma with squamous metaplasia of the gallbladder; squamous cell carcinoma of the gallbladder; adenocarcinoma of the extrahepatic bile duct; cholangiocarcinoma of the gallbladder; cholangiocarcinoma of the extrahepatic bile duct
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — Capecitabine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Capecitabine + Gemcitabine (Experimental): Capecitabine 650 mg/m^2 twice daily (BID), by mouth (PO) at 12 hour intervals, Days 1-14, every 21 days; Gemcitabine 1000 mg/m^2, intravenous (IV) over 100 minutes, Days 1, 8, every 21 days
  Interventions: Drug: capecitabine; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: capecitabine — 650 mg/m^2 twice daily (BID), by mouth (PO) at 12 hour intervals, Days 1-14, every 21 days
  Other Names: Xeloda (NSC-712807)
Drug: gemcitabine hydrochloride — 1000 mg/m^2, intravenous (IV) over 100 minutes, Days 1,8, every 21 days
  Other Names: Gemzar (NSC-613327)

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and capecitabine, use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining gemcitabine with capecitabine in treating patients who have locally advanced or metastatic gallbladder cancer or cholangiocarcinoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rates (confirmed complete and partial responses) in patients with unresectable, locally advanced or metastatic gallbladder cancer or cholangiocarcinoma treated with gemcitabine and capecitabine.
* Determine the overall survival of patients treated with this regimen.
* Determine the quantitative and qualitative toxic effects of this regimen in these patients.
* Determine the feasibility of accruing patients with these disease sites.
* Evaluate, preliminarily, relevant prognostic markers in these disease sites and the prognostic implications as predictors of survival in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive oral capecitabine twice daily on days 1-14 and gemcitabine IV over 100 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months until disease progression and then every 6 months for up to 3 years.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study within approximately 10-20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed gallbladder cancer or cholangiocarcinoma

  * Locally advanced or metastatic disease that is unresectable
  * Eligible subtypes:

    * Adenocarcinoma, intestinal type
    * Adenocarcinoma, not otherwise specified (NOS)
    * Papillary carcinoma
    * Clear cell adenocarcinoma
    * Mucinous carcinoma
    * Signet ring cell carcinoma
    * Squamous cell carcinoma
    * Adenosquamous carcinoma
    * Small cell carcinoma
    * Undifferentiated carcinoma
    * Carcinoma, NOS

OR

* Histologically confirmed adenocarcinoma of a metastatic site with clinical documentation* of gallbladder or bile duct involvement and no evidence of another primary

NOTE: *If clinical documentation of gallbladder or bile duct involvement is not possible due to removal of the organ, a clinically and/or radiographically consistent picture plus pathologic findings from the metastatic site consistent with cholangiocarcinoma are allowed

* Measurable disease located outside prior radiotherapy port
* No carcinoid tumors or sarcomas

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 3 times upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) or Serum glutamic pyruvic transaminase (SGPT) no greater than 2.5 times ULN (5 times ULN if liver metastasis is present)

Renal:

* Creatinine clearance at least 30 mL/min

Cardiovascular:

* No clinically significant cardiac disease that is not well controlled by medication
* No congestive heart failure
* No symptomatic coronary artery disease
* No cardiac arrhythmias
* No myocardial infarction within the past 12 months

Gastrointestinal:

* Able to swallow and/or receive medications via gastrostomy feeding tube
* No intractable nausea or vomiting
* No malabsorption syndrome

Other:

* No severe reaction to fluoropyrimidine therapy or known hypersensitivity to fluorouracil
* No other malignancy within the past 5 years except:

  * Adequately treated basal cell or squamous cell skin cancer
  * Carcinoma in situ of the cervix
  * Adequately treated stage I or II cancer currently in complete remission
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior neoadjuvant or adjuvant immunotherapy allowed provided therapy was completed at least 1 year before documented recurrence or metastatic disease
* No concurrent immunotherapy

Chemotherapy:

* Prior neoadjuvant or adjuvant chemotherapy or chemoradiotherapy allowed provided therapy was completed at least 1 year before documented recurrence or metastatic disease
* No other concurrent chemotherapy

Endocrine therapy:

* Prior neoadjuvant or adjuvant hormonal therapy allowed provided therapy was completed at least 1 year before documented recurrence or metastatic disease
* No concurrent hormonal therapy

Radiotherapy:

* See Disease Characteristics
* See Chemotherapy
* Recovered from prior radiotherapy
* Prior neoadjuvant or adjuvant radiotherapy allowed provided therapy was completed at least 1 year before documented recurrence or metastatic disease
* No prior radiotherapy to 25% or more of bone marrow
* No concurrent radiotherapy except for palliation of metastatic sites not considered target lesions

Surgery:

* At least 2 weeks since prior surgery for this malignancy and recovered

Other:

* No prior treatment for metastatic disease
* No other concurrent therapy for this cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2003-09; Primary Completion 2008-04 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Syma Iqbal, MD, Study Chair — University of Southern California; Heinz-Josef Lenz, MD, Study Chair — University of Southern California
Locations (112):
- United States (112):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - North Bay Cancer Center, Fairfield, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - West Florida Regional Medical Center, Pensacola, Florida
  - Hematology Oncology Associates of Eastern Idaho, Idaho Falls, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Cancer Care Center at St. Francis Hospital, Indianapolis, Indiana
  - South Central Kansas Regional Medical Center, Arkansas City, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Pratt Cancer Center of Kansas, Pratt, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates in Womens Health, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Louisiana State University Health Sciences Center - Monroe, Monroe, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Cancer Treatment Center at Christus Schumpert St. Mary Place, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Cancer Center at Thibodaux Regional Medical Center, Thibodaux, Louisiana
  - Battle Creek Health System, Battle Creek, Michigan
  - Mecosta County General Hospital, Big Rapids, Michigan
  - Josephine Ford Cancer Center at Henry Ford Health System, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Mercy Medical Center, Grand Rapids, Michigan
  - Spectrum Health Cancer Care - Butterworth Campus, Grand Rapids, Michigan
  - Metropolitan Hospital, Grand Rapids, Michigan
  - Spectrum Health Hospital - Blodgett Campus, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Cape Girardeau, Missouri
  - St. Francis Medical Center, Cape Girardeau, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute, Great Falls, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - Adirondack Cancer Care, Glens Falls, New York
  - Orange Regional Medical Center - Horton Campus, Middletown, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Cancer Center at Iredell Memorial Hospital, Statesville, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - University Hospitals Ireland Cancer Center at Mercy Medical Center, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Oncology Group - Independence, Independence, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Veterans Affairs Medical Center - Amarillo, Amarillo, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Memorial Hospital of Martinsville and Henry County, Martinsville, Virginia
  - St. Joseph Hospital Community Cancer Center, Bellingham, Washington
  - Harborview Medical Center, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Central Washington Hospital, Wenatchee, Washington
  - Wenatchee Valley Clinic, Wenatchee, Washington

REFERENCES:
- [Background] Lurje G, Zhang W, Yang D, Groshen S, Hendifar AE, Husain H, Nagashima F, Chang HM, Fazzone W, Ladner RD, Pohl A, Ning Y, Iqbal S, El-Khoueiry A, Lenz HJ. Thymidylate synthase haplotype is associated with tumor recurrence in stage II and stage III colon cancer. Pharmacogenet Genomics. 2008 Feb;18(2):161-8. doi: 10.1097/FPC.0b013e3282f4aea6. PMID 18192902
- [Result] Iqbal S, Rankin C, Lenz HJ, Gold PJ, Ahmad SA, El-Khoueiry AB, Messino MJ, Holcombe RF, Blanke CD. A phase II trial of gemcitabine and capecitabine in patients with unresectable or metastatic gallbladder cancer or cholangiocarcinoma: Southwest Oncology Group study S0202. Cancer Chemother Pharmacol. 2011 Dec;68(6):1595-602. doi: 10.1007/s00280-011-1657-1. Epub 2011 May 10. PMID 21556747

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Capecitabine + Gemcitabine
Started | 57
Eligible | 54
Eligible and Began Protocol Therapy | 52 (One patient went off study prior to any toxicity assessments and is not evaluable for toxicities.)
Completed | 0
Not Completed | 57
Not completed — Adverse Event | 14
Not completed — Death | 1
Not completed — Progression | 26
Not completed — Withdrawal by Subject | 6
Not completed — Other | 5
Not completed — Ineligible | 3
Not completed — Never received treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | Capecitabine + Gemcitabine
Number analyzed (Participants) | 52
Age, Continuous [Median (Full Range); unit: years] | 58.8 [29.5 to 85.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 37
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Response
Description: Complete Response (CR) is complete disappearance of all measurable and non-measurable disease. No new lesions, no disease related symptoms. Normalization of markers and other abnormal lab values. Partial Response (PR) is greater than or equal to 30% decrease under baseline of the sum of longest diameters of all target measurable lesions. No unequivocal progression of non-measurable disease. No new lesions. Confirmation of CR or PR means a repeat scan at least 4 weeks apart documented before progression or symptomatic deterioration. Progression is 20% increase in sum of longest diameters of target measurable lesions over smallest sum observed and/or unequivocal progression of non-measurable disease and/or appearance of new lesion/site or death due to disease without prior documentation of progression and without symptomatic deterioration. Symptomatic deterioration is global deterioration of health status requiring discontinuation of treatment without objective evidence of progression.
Time Frame: Patients assessed at least every six weeks while on protocol treatment
Population: All eligible patients who started treatment were included in assessing response estimates.
Measure: Number; unit: participants
Arm/Group | Capecitabine + Gemcitabine
Number analyzed (Participants) | 52
participants
  Confirmed Partial Response | 7
  Unconfirmed Partial Response | 6
  Stable Disease | 12
  Progression | 15
  Symptomatic Deterioration | 3
  Early Death | 1
  Inadequate Assessment | 8

2. Secondary Outcome: Overall Survival
Description: Measured from time of registration to death, or last contact date
Time Frame: All patients will be followed until death or three years after registration, whichever is first.
Population: All eligible patients who started treatment were included in assessing response estimates.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capecitabine + Gemcitabine
Number analyzed (Participants) | 52
months | 7 [5 to 8]

3. Secondary Outcome: Number of Patients With Grade 3 Through 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0. Any CTCAE 3.0 event of Grade 3 (severe), Grade 4 (life threatening) or Grade 5 (fatal) which were deemed to be related to protocol treatment are included. For each patient, worst grade of each event type is reported.
Time Frame: Patients were assessed for adverse events 3 weeks after starting treatment. Assessments for adverse events continued every 3 weeks for the duration of protocol treatment.
Population: Eligible patients who received any treatment and were assessed for toxicity were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (severe), Grade 4 (life threatening) or Grade 5 (fatal) which were deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Groups:
- Gemcitabine and Capecitabine: Capecitabine 650 mg/m^2 twice daily (BID), by mouth (PO) at 12 hour intervals, Days 1-14, every 21 days; Gemcitabine 1000 mg/m^2, intravenous (IV) over 100 minutes, Days 1, 8, every 21 days
Arm/Group | Gemcitabine and Capecitabine
Number analyzed (Participants) | 51
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 1
  AST,SGOT (serum glutamic oxaloacetic transaminase) | 5
  Albumin, serum-low (hypoalbuminemia) | 1
  Alkaline phosphatase | 5
  Anorexia | 2
  Ascites (non-malignant) | 1
  Bilirubin (hyperbilirubinemia) | 4
  Constipation | 1
  Creatinine | 1
  Dehydration | 3
  Diarrhea | 1
  Dysphagia (difficulty swallowing) | 1
  Fatigue (asthenia, lethargy, malaise) | 8
  Hemoglobin | 6
  Hemolysis | 1
  Hemorrhage, GI - Esophagus | 1
  Infection w/Grade 3-4 neutrophils - Upper airway | 1
  Infection with normal ANC or Grade 1-2 neutrophils | 1
  Leukocytes (total WBC) | 9
  Mucositis/stomatitis (clinical exam) - Oral cavity | 1
  Mucositis/stomatitis (function/symp)-Oral cavity | 1
  Muscle weakness (not due to neuropathy) | 1
  Nausea | 3
  Neutrophils/granulocytes (ANC/AGC) | 16
  Pain - Abdomen NOS | 2
  Pain - Joint | 1
  Pain - Muscle | 1
  Pain - Tumor pain | 1
  Platelets | 12
  Potassium, serum-low (hypokalemia) | 2
  Rash: hand-foot skin reaction | 4
  Supraventricular nodal arrhythmia | 1
  Thrombosis/thrombus/embolism | 1
  Vomiting | 2

4. Secondary Outcome: Accrual of Patients With This Disease Site
Description: Only eligible patients who received treatment were evaluable for response and survival outcomes.
Time Frame: 1-20 months
Population: Patients with advanced disease accrued between September 2003 to April 2005
Measure: Number; unit: participants
Arm/Group | Capecitabine + Gemcitabine
Number analyzed (Participants) | 57
participants
  Eligible | 54
  Eligible and Analyzable | 52

5. Secondary Outcome: Median Survival Time for Participants With Relevant Biologic Markers
Description: To evaluate in a preliminary fashion relevant prognostic markers in gallbladder and cholangiocarcinoma which may have prognostic implications as predictors of survival. Overall survival measured from time of registration to death, or last contact date.
Time Frame: All patients will be followed until death or three years after registration, whichever is first.
Population: Eligible patients who received genotyping were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capecitabine + Gemcitabine
Number analyzed (Participants) | 22
months
  TS 3' +/+ (N=14) | 7 [4 to 13]
  TS 3' +/- (N=6) | 7 [2 to 7]
  TS 3' -/- (N=2) | 9 [2 to NA] — insufficient number of participants
  TS 5' Low functional significance (N=16) | 9 [4 to 12]
  TS 5' Intermediate functional significance (N=16) | 7 [2 to 7]
  MTHFR C677T - C/C (N=11) | 6 [4 to 9]
  MTHFR C677T - C/T (N=11) | 7 [2 to 13]
  MTHFR A1298C - A/A (N=11) | 7 [4 to 12]
  MTHFR A1298C - A/C (N=8) | 4 [2 to 6]
  MTHFR A1298C - C/C (N=3) | 9 [5 to 9]
  RRMI G/A - G/G (N=9) | 7 [4 to 7]
  RRMI G/A - G/A (N=10) | 9 [2 to 12]
  RRMI G/A - A/A (N=3) | 5 [4 to 5]
  CDA A79C - A/A (N=8) | 4 [2 to 5]
  CDA A79C - A/C (N=12) | 7 [5 to 9]
  CDA A79C - C/C (N=1) | NA [NA to NA] — insufficient number of participants

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events 3 weeks after starting treatment. Assessments for adverse events continued every 3 weeks for the duration of protocol treatment.
Description: One patient went off study prior to any toxicity assessments and is not evaluable for toxicities.
Arm/Group | Gemcitabine and Capecitabine
Serious Adverse Events (participants affected / at risk) | 7/51
Other Adverse Events (participants affected / at risk) | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine and Capecitabine (N=51)
Constitutional Symptoms-Other (Specify) (General disorders) | 2 — Death - progressive disease
Hepatobiliary/Pancreas-Biliary obstruction (Hepatobiliary disorders) | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Blood (Infections and infestations) | 1
Bilirubin (hyperbilirubinemia) (Investigations) | 1
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine and Capecitabine (N=51)
Hemoglobin (Blood and lymphatic system disorders) | 42
Ocular surface disease (Eye disorders) | 3
Ascites (non-malignant) (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 21
Diarrhea (Gastrointestinal disorders) | 17
Heartburn/dyspepsia (Gastrointestinal disorders) | 4
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 11
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 32
Pain - Abdomen NOS (Gastrointestinal disorders) | 18
Vomiting (Gastrointestinal disorders) | 19
Edema: limb (General disorders) | 12
Fatigue (asthenia, lethargy, malaise) (General disorders) | 44
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 15
Injection site reaction/extravasation changes (General disorders) | 3
Pain-Other (Specify) (General disorders) | 4
Rigors/chills (General disorders) | 10
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 7
Inf w/normal ANC or Gr 1-2 neutrophils - Bladder (Infections and infestations) | 4
Inf w/normal ANC or Gr 1-2 neutrophils - Skin (Infections and infestations) | 3
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 12
AST, SGOT (Investigations) | 39
Alkaline phosphatase (Investigations) | 36
Bilirubin (hyperbilirubinemia) (Investigations) | 13
Creatinine (Investigations) | 3
GGT (gamma-glutamyl transpeptidase) (Investigations) | 3
Leukocytes (total WBC) (Investigations) | 29
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 30
Platelets (Investigations) | 29
Weight loss (Investigations) | 8
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 13
Anorexia (Metabolism and nutrition disorders) | 14
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 4
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 18
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 3
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 5
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 9
Muscle weakness, not d/t neuropathy - Extrem-lower (Musculoskeletal and connective tissue disorders) | 3
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 3
Pain - Back (Musculoskeletal and connective tissue disorders) | 8
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 3
Pain - Joint (Musculoskeletal and connective tissue disorders) | 4
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 4
Pain - Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14
Neuropathy: sensory (Nervous system disorders) | 5
Pain - Head/headache (Nervous system disorders) | 7
Taste alteration (dysgeusia) (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 5
Mood alteration - anxiety (Psychiatric disorders) | 4
Mood alteration - depression (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 13
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 12
Nail changes (Skin and subcutaneous tissue disorders) | 6
Pruritus/itching (Skin and subcutaneous tissue disorders) | 10
Rash/desquamation (Skin and subcutaneous tissue disorders) | 14
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 11
Thrombosis/thrombus/embolism (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No